CLINICAL TRIAL: NCT00794118
Title: Drug Outcome Survey for Biological Treatments in Rheumatoid Arthritis: an Observational Study
Brief Title: Drug Outcome Survey for Biological Treatments in Rheumatoid Arthritis: an Observational Study (Dose)
Acronym: DOSE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A1-102321; B1801119
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2012-05-16 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1.0: As per routinary clinical practice
  Interventions: Other: As per clinical practice

INTERVENTIONS:
Other: As per clinical practice — As per clinical practice
  Other Names: Observational study

SUMMARY:
The primary purpose of this observational study is to describe and define the current daily practice of management of anti-TNF-agents in Rheumatoid Arthritis (RA) patients. Data will be collected only from subjects providing informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older
2. Diagnosis of RA in accordance with ARA 1987 classification has satisfied at least 4 of the following 7 criteria:

   1. Morning stiffness in and around the joints lasting at least 1 hour;
   2. Arthritis of 3 or more joint areas;
   3. Arthritis of hand joints;
   4. Symmetric arthritis. simultaneous involvement of the same joint areas on both sides of the body;
   5. Rheumatoid nodules;
   6. Serum Rheumatoid Factor (RF)
   7. Radiographic changes. Criteria 1 through 4 must have been present for at least 6 weeks.
3. Patients refractory or without complete response to DMARDs according to the Italian Guidelines for the clinical practice established by Italian Society of Rheumatology
4. Patients naive to anti-TNF drugs
5. Outpatients

Exclusion Criteria:

Patients involved in controlled or interventional trials in the 12 previous months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Roma, Italy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-102321&StudyName=Drug%20Outcome%20Survey%20for%20Biological%20Treatments%20in%20Rheumatoid%20Arthritis%3A%20an%20Observational%20Study%20%28Dose%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-tumor Necrosis Factor (Anti-TNF) Agents: Participants with rheumatoid arthritis (RA) prescribed with anti-TNF agents (etanercept, adalimumab, infliximab) as per investigator's discretion were observed for a period of 12 months.
Period: Overall Study
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Started | 299
Completed | 272
Not Completed | 27
Not completed — Lost to Follow-up | 16
Not completed — Withdrawal by Subject | 9
Not completed — Changed hospital center | 2

BASELINE CHARACTERISTICS:
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 299
Age, Customized [Number; unit: Participants]
  18 to 34 years | 29
  35 to 49 years | 72
  50 to 64 years | 133
  Greater than or equal to (>=) 65 years | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230
  Male | 69
Percentage of participants with Disease Activity Score Based on 28-joints count (DAS28) remission [Number; unit: Percentage of participants] — DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the ESR and PtGA of disease activity. DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity. A participant is considered to be in remission if they have a DAS28 <2.6.
  Percentage of participants | 1.7
Disease Activity Score Based on 28-joints count (DAS28) [Mean (Standard Deviation); unit: Units on a scale] — DAS28 calculated from the SJC and PJC using the 28 joints count, the ESR and PtGA of disease activity. DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity. Number of participants analyzed (N)=272 for this parameter.
  Units on a scale | 5.4 (1.2)
Patient Global Assessment (PtGA) [Mean (Standard Deviation); unit: centimeter (cm)] — PtGA measured using a 10 cm Visual Analog Scale (VAS) ranging from 0 cm = very good to 10 cm = very bad.
  centimeter (cm) | 6.6 (2.1)
Physician Global Assessment (PGA) [Mean (Standard Deviation); unit: cm] — PGA was measured on a 0 to 10 cm VAS, with 0 cm = no disease activity to 10 cm = worst disease activity possible.
  cm | 6.1 (1.7)
Visual Analogue Scale for Pain (VAS-pain) [Mean (Standard Deviation); unit: cm] — 10 cm line (VAS) marked by participant. Intensity of pain range: 0 cm = no pain to 10 cm = worst possible pain.
  cm | 6.7 (2.2)
C-reactive Protein (CRP) [Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)] — CRP is a marker of inflammation. CRP value higher than 0.5 mg/dL is consistent with inflammation. Number of participants analyzed (N) = 272 for this parameter.
  milligram/deciliter (mg/dL) | 3.3 (6.3)
Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: millimeter/hour (mm/hr)] — ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A higher rate is consistent with inflammation.
  millimeter/hour (mm/hr) | 32.9 (22.0)
Rheumatoid Factor (RF) [Number; unit: Participants] — RF is the auto antibody directed against immunoglobulin G (IgG) and its concentration is observed in human serum or plasma. RF value higher than 20 unit/milliliter (U/mL) is considered positive.
  Participants
    Positive | 163
    Negative | 118
    Not available (NA) | 18
Anti-cyclic Citrullinated Protein (Anti-CCP) antibodies [Number; unit: Participants] — Anti-CCP antibodies are auto antibodies (antibodies directed against 1 or more of an individual's own proteins) that are frequently detected in the blood of rheumatoid arthritis participants. Anti-CCP antibodies value higher than 10 U/mL is considered positive.
  Participants
    Positive | 124
    Negative | 97
    NA | 78
Anti-nuclear antibodies [Number; unit: Participants] — Anti-nuclear antibodies are auto antibodies directed against contents of the nucleus and are present in higher than normal numbers in autoimmune disease. Anti-nuclear antibodies value higher than 1:160 is considered positive.
  Participants
    Positive | 38
    Negative | 170
    NA | 91
Anti-deoxyribonucleic Acid (Anti-DNA) antibodies [Number; unit: Participants] — Anti-DNA antibodies are auto antibodies directed against DNA and are present in higher than normal numbers in autoimmune disease. Anti-DNA antibodies value higher than 1:20 is considered positive.
  Participants
    Positive | 6
    Negative | 173
    NA | 120
Duration of morning stiffness [Mean (Standard Deviation); unit: minutes] — Duration of morning stiffness: Time elapsed when participant woke up in morning and was able to resume normal activities without stiffness in minutes. Increase in stiffness duration from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
  minutes | 61.8 (48.0)
Stanford Health Assessment Questionnaire (HAQ) [Mean (Standard Deviation); unit: Units on a scale] — HAQ is a measure of functional limitations. Participants were rated on 4 point scale with scores: 0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do based on degree of difficulty experienced with 20 tasks grouped into 8 areas of dressing, rising, hygiene, reach, walking, eating, grip and activities. Average score range: 0 to 3.
  Units on a scale | 1.4 (0.7)
36-Item Short-Form Health Survey (SF-36) [Mean (Standard Deviation); unit: Units on a Scale] — SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
  Units on a Scale
    Indice sintetico salute fisica del (ISF) | 38.8 (10.6)
    Indice sintetico salute mentale del (ISM) | 48.0 (13.2)
Disease duration [Median (Inter-Quartile Range); unit: Years] | 5.0 [2.0 to 10.0]
Number of tender joints [Mean (Standard Deviation); unit: Tender joints] — The mean number of tender joints was evaluated based on the number of tender joints in a standard 28 joint count.
  Tender joints | 11.0 (7.1)
Number of swollen joints (SJC) [Mean (Standard Deviation); unit: Swollen joints] — The mean number of swollen joints was evaluated based on the number of swollen joints in a standard 28 joint count.
  Swollen joints | 7.3 (5.3)
Percentage of participants given Disease Modifying Anti-Rheumatoid Drugs (DMARD) [Number; unit: Percentage of participants] | 98.3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Activity Score Based on 28-joints Count (DAS28) Remission at Month 3
Description: DAS28 calculated from the SJC and PJC using the 28 joints count, the ESR (mm/hr) and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 less than or equal to (<=) 3.2 = low disease activity, DAS28 greater than (>) 3.2 to 5.1 = moderate to high disease activity. A participant is considered to be in remission if they have a DAS28 less than (<) 2.6.
Time Frame: Month 3
Population: Intent-to-Treat (ITT) population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Percentage of participants | 13.4

2. Primary Outcome: Percentage of Participants With Disease Activity Score Based on 28-joints Count (DAS28) Remission at Month 6
Description: DAS28 calculated from the SJC and PJC using the 28 joints count, the ESR (mm/hr) and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity. A participant is considered to be in remission if they have a DAS28 <2.6.
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Percentage of participants | 21.6

3. Primary Outcome: Percentage of Participants With Disease Activity Score Based on 28-joints Count (DAS28) Remission at Month 9
Description: as for outcome 2
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Percentage of participants | 27.2

4. Primary Outcome: Percentage of Participants With Disease Activity Score Based on 28-joints Count (DAS28) Remission at Month 12
Description: DAS28 calculated from the SJC and PJC using the 28 joints count, the ESR (mm/hr) and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity. A participant is considered to be in remission if they have a DAS28 < 2.6.
Time Frame: Month 12
Population: ITT population included all participants who received at least 1 dose of the study medication. Missing values were imputed using last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Percentage of participants | 22.6

5. Primary Outcome: Disease Activity Score Based on 28-joints Count (DAS28) at Month 3
Description: DAS28 calculated from the SJC and PJC using the 28 joints count, the ESR (mm/hr) and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Units on a Scale | 4.2 (1.3)

6. Primary Outcome: Disease Activity Score Based on 28-joints Count (DAS28) at Month 6
Description: as for outcome 5
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Units on a Scale | 3.7 (1.3)

7. Primary Outcome: Disease Activity Score Based on 28-joints Count (DAS28) at Month 9
Description: as for outcome 5
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Units on a Scale | 3.4 (1.2)

8. Primary Outcome: Disease Activity Score Based on 28-joints Count (DAS28) at Month 12
Description: as for outcome 5
Time Frame: Month 12
Population: ITT population included all participants who received at least 1 dose of the study medication. Missing values were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Units on a Scale | 3.6 (1.5)

9. Primary Outcome: Patient Global Assessment (PtGA) of Disease Activity Score at Month 3
Description: PtGA measured using a 10 cm (VAS) ranging from 0 cm = very good to 10 cm = very bad.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 4.1 (2.3)

10. Primary Outcome: Patient Global Assessment (PtGA) of Disease Activity Score at Month 6
Description: PtGA measured using a 10 cm (VAS) ranging from 0 cm = very good to 10 cm = very bad.
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 3.4 (2.4)

11. Primary Outcome: Patient Global Assessment (PtGA) of Disease Activity Score at Month 9
Description: PtGA measured using a 10 cm (VAS) ranging from 0 cm = very good to 10 cm = very bad.
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 2.8 (2.3)

12. Primary Outcome: Patient Global Assessment (PtGA) of Disease Activity Score at Month 12
Description: PtGA measured using a 10 cm (VAS) ranging from 0 cm = very good to 10 cm = very bad.
Time Frame: Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 3.3 (2.6)

13. Primary Outcome: Physician Global Assessment (PGA) of Disease Activity at Month 3
Description: PGA was measured on a 0 to 10 cm VAS, with 0 cm = no disease activity to 10 cm = worst disease activity possible.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 3.7 (2.1)

14. Primary Outcome: Physician Global Assessment (PGA) of Disease Activity at Month 6
Description: PGA was measured on a 0 to 10 cm VAS, with 0 cm = no disease activity to 10 cm = worst disease activity possible.
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 2.9 (2.1)

15. Primary Outcome: Physician Global Assessment (PGA) of Disease Activity at Month 9
Description: PGA was measured on a 0 to 10 cm VAS, with 0 cm = no disease activity to 10 cm = worst disease activity possible.
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 2.3 (2.1)

16. Primary Outcome: Physician Global Assessment (PGA) of Disease Activity at Month 12
Description: PGA was measured on a 0 to 10 cm VAS, with 0 cm = no disease activity to 10 cm = worst disease activity possible.
Time Frame: Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 2.8 (2.4)

17. Primary Outcome: Visual Analogue Scale for Pain (VAS-pain) at Month 3
Description: 10 cm line (VAS) marked by participant. Intensity of pain range 0 cm = no pain to 10 cm = worst possible pain.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 4.1 (2.4)

18. Primary Outcome: Visual Analogue Scale for Pain (VAS-pain) at Month 6
Description: 10 cm line (VAS) marked by participant. Intensity of pain range 0 cm = no pain to 10 cm = worst possible pain.
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 3.3 (2.3)

19. Primary Outcome: Visual Analogue Scale for Pain (VAS-pain) at Month 9
Description: 10 cm line (VAS) marked by participant. Intensity of pain range 0 cm = no pain to 10 cm = worst possible pain.
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 2.9 (2.4)

20. Primary Outcome: Visual Analogue Scale for Pain (VAS-pain) at Month 12
Description: 10 cm line (VAS) marked by participant. Intensity of pain range 0 cm = no pain to 10 cm = worst possible pain.
Time Frame: Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
cm | 3.3 (2.7)

21. Primary Outcome: C-reactive Protein (CRP) at Month 3
Description: CRP is a marker of inflammation. CRP value higher than 0.5 mg/dL is consistent with inflammation.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
mg/dL | 1.4 (2.5)

22. Primary Outcome: C-reactive Protein (CRP) at Month 6
Description: CRP is a marker of inflammation. CRP value higher than 0.5 mg/dL is consistent with inflammation.
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
mg/dL | 1.3 (2.5)

23. Primary Outcome: C-reactive Protein (CRP) at Month 9
Description: CRP is a marker of inflammation. CRP value higher than 0.5 mg/dL is consistent with inflammation.
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
mg/dL | 1.1 (1.6)

24. Primary Outcome: C-reactive Protein (CRP) at Month 12
Description: CRP is a marker of inflammation. CRP value higher than 0.5 mg/dL is consistent with inflammation.
Time Frame: Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
mg/dL | 1.5 (2.6)

25. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) at Month 3
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A higher rate is consistent with inflammation.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
mm/hr | 23.9 (18.8)

26. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) at Month 6
Description: as for outcome 25
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
mm/hr | 20.8 (16.2)

27. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) at Month 9
Description: as for outcome 25
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
mm/hr | 18.4 (13.5)

28. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) at Month 12
Description: as for outcome 25
Time Frame: Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
mm/hr | 21.9 (18.9)

29. Primary Outcome: Number of Participants With Rheumatoid Factor (RF) at Month 3
Description: RF is the auto antibody directed against IgG and its concentration is observed in human serum or plasma. RF value higher than 20 U/mL is considered positive.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 80
  Negative | 88
  NA | 98

30. Primary Outcome: Number of Participants With Rheumatoid Factor (RF) at Month 6
Description: as for outcome 29
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 77
  Negative | 74
  NA | 83

31. Primary Outcome: Number of Participants With Rheumatoid Factor (RF) at Month 9
Description: as for outcome 29
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 63
  Negative | 57
  NA | 106

32. Primary Outcome: Number of Participants With Rheumatoid Factor (RF) at Month 12
Description: as for outcome 29
Time Frame: Month 12
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 88
  Negative | 67
  NA | 117

33. Primary Outcome: Number of Participants With Anti-cyclic Citrullinated Protein (Anti-CCP) Antibodies at Month 3
Description: Anti-CCP antibodies are auto antibodies (antibodies directed against 1 or more of an individual's own proteins) that are frequently detected in the blood of rheumatoid arthritis participants. Anti-CCP antibodies value higher than 10 U/mL is considered positive.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 43
  Negative | 50
  NA | 174

34. Primary Outcome: Number of Participants With Anti-cyclic Citrullinated Protein (Anti-CCP) Antibodies at Month 6
Description: as for outcome 33
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 44
  Negative | 44
  NA | 147

35. Primary Outcome: Number of Participants With Anti-cyclic Citrullinated Protein (Anti-CCP) Antibodies at Month 9
Description: as for outcome 33
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 32
  Negative | 39
  NA | 154

36. Primary Outcome: Number of Participants With Anti-cyclic Citrullinated Protein (Anti-CCP) Antibodies at Month 12
Description: as for outcome 33
Time Frame: Month 12
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 52
  Negative | 45
  NA | 175

37. Primary Outcome: Number of Participants With Anti-nuclear Antibodies at Month 3
Description: Anti-nuclear antibodies are auto antibodies directed against contents of the nucleus and are present in higher than normal numbers in autoimmune disease. Anti-nuclear antibodies value higher than 1:160 is considered positive.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 8
  Negative | 78
  NA | 181

38. Primary Outcome: Number of Participants With Anti-nuclear Antibodies at Month 6
Description: as for outcome 37
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 14
  Negative | 79
  NA | 142

39. Primary Outcome: Number of Participants With Anti-nuclear Antibodies at Month 9
Description: as for outcome 37
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 9
  Negative | 57
  NA | 159

40. Primary Outcome: Number of Participants With Anti-nuclear Antibodies at Month 12
Description: as for outcome 37
Time Frame: Month 12
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 14
  Negative | 85
  NA | 173

41. Primary Outcome: Number of Participants With Anti-deoxyribonucleic Acid (Anti-DNA) Antibodies at Month 3
Description: Anti-DNA antibodies are auto antibodies directed against DNA and are present in higher than normal numbers in autoimmune disease. Anti-DNA antibodies value higher than 1:20 is considered positive.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 1
  Negative | 79
  NA | 187

42. Primary Outcome: Number of Participants With Anti-deoxyribonucleic Acid (Anti-DNA) Antibodies at Month 6
Description: as for outcome 41
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 1
  Negative | 80
  NA | 154

43. Primary Outcome: Number of Participants With Anti-deoxyribonucleic Acid (Anti-DNA) Antibodies at Month 9
Description: as for outcome 41
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 4
  Negative | 60
  NA | 161

44. Primary Outcome: Number of Participants With Anti-deoxyribonucleic Acid (Anti-DNA) Antibodies at Month 12
Description: as for outcome 41
Time Frame: Month 12
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Participants
  Positive | 3
  Negative | 88
  NA | 181

45. Primary Outcome: Duration of Morning Stiffness at Month 3
Description: Duration of morning stiffness: Time elapsed when participant woke up in morning and was able to resume normal activities without stiffness in minutes. Increase in stiffness duration from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
minutes | 26.4 (26.3)

46. Primary Outcome: Duration of Morning Stiffness at Month 6
Description: as for outcome 45
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
minutes | 19.6 (32.7)

47. Primary Outcome: Duration of Morning Stiffness at Month 9
Description: as for outcome 45
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
minutes | 13.2 (17.5)

48. Primary Outcome: Duration of Morning Stiffness at Month 12
Description: as for outcome 45
Time Frame: Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
minutes | 17.8 (23.8)

49. Primary Outcome: Stanford Health Assessment Questionnaire (HAQ) Score at Month 3
Description: HAQ is a measure of functional limitations. Participants were rated on 4 point scale with scores: 0=no difficulty (normal), 1=some difficulty (adequate), 2=much difficulty (limited), 3=unable to do based on degree of difficulty experienced with 20 tasks grouped into 8 areas of dressing, rising, hygiene, reach, walking, eating, grip and activities. The higher score reported by the participant for any component question of the 8 categories determines the score for that categories. Total score is divided for 8. Average score range: 0 (no difficulty) to 3 (unable to do).
Time Frame: Month 3
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Units on a Scale | 1.0 (0.7)

50. Primary Outcome: Stanford Health Assessment Questionnaire (HAQ) Score at Month 6
Description: as for outcome 49
Time Frame: Month 6
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Units on a Scale | 0.7 (0.7)

51. Primary Outcome: Stanford Health Assessment Questionnaire (HAQ) Score at Month 9
Description: as for outcome 49
Time Frame: Month 9
Population: ITT population included all participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Units on a Scale | 0.7 (0.7)

52. Primary Outcome: Stanford Health Assessment Questionnaire (HAQ) Score at Month 12
Description: as for outcome 49
Time Frame: Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Units on a Scale | 0.8 (0.7)

53. Primary Outcome: 36-Item Short-Form Health Survey (SF-36) at Month 12
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Month 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 272
Units on a Scale
  ISF | 52.2 (14.7)
  ISM | 55.5 (11.8)

54. Secondary Outcome: Direct Costs
Description: Direct costs included all expenses requiring actual payment or time spent due to the disease itself or to disability.
Time Frame: Baseline, Months 3, 6, 9 and 12
Population: There was not a direct data collection on costs. Zero participants were analyzed for this outcome measure.
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 0

55. Secondary Outcome: Indirect Costs
Description: Indirect costs represent the loss of resources as a consequence of work disability or unemployment.
Time Frame: Baseline, Months 3, 6, 9 and 12
Population: There was not a direct data collection on costs. Zero participants were analyzed for this outcome measure.
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Anti-tumor Necrosis Factor (Anti-TNF) Agents
Serious Adverse Events (participants affected / at risk) | 0/272
Other Adverse Events (participants affected / at risk) | 21/272
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-tumor Necrosis Factor (Anti-TNF) Agents (N=272)
Infusion related reaction (Immune system disorders) | 13
Bronchopulmonary infection (Respiratory, thoracic and mediastinal disorders) | 3
Injection site reaction (General disorders) | 2
Blood pressure high (Vascular disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Protocol did not indicate primary or secondary endpoints and all determination of primary or secondary endpoints were arbitrary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.